CLINICAL TRIAL: NCT04786184
Title: Capnography-Assisted Learned Monitored (CALM) Breathing Therapy for COPD
Acronym: CALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAT8556; 20-00751 (Other: NYU Langone Health); R34AT010673 (NIH)
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: COPD
Keywords: Breathing; Anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A prospective RCT: In Phase I, participants will be randomized 1:1 to one of two groups: CALM Breathing (N = 25) and Wait-List control (N = 25). In Phase II, both groups will be offered Columbia University's 10-week PR program (care as usual). Access to timely initiation of PR will be facilitated. We will use a hybrid design to evaluate feasibility and acceptability.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALM Breathing (Experimental)
  Interventions: Behavioral: CALM Breathing
- Wait-List Control (Active Comparator)
  Interventions: Behavioral: Traditional outpatient PR

INTERVENTIONS:
Behavioral: CALM Breathing — CALM Breathing is a mind-body breathing therapy that links CO2 changes to dyspnea and anxiety symptoms and targets breathing efficiency and self-efficacy in COPD. CALM Breathing: Individual interoception- based breathing therapy with capnography (non- exercise training) Home Program: Monitored home- based breathing exercises; RR biofeedback; goal setting; exercise logging. Coaching: Motivational interviewing. Personnel: PT, EP, occupational therapist, or nurse. Frequency: 1-hour sessions, twice per week for 4 weeks. Exercises: • 10 core breathing exercises with ETCO2 biofeedback in recovery postures at rest and with body movement (gentle stretches and brief low-moderate intensity physical activity). • Breathing biofeedback (ETCO2, RR, airflow pattern). Education: Education on anxiety; COPD Patient Guide.
  Arms: CALM Breathing
Behavioral: Traditional outpatient PR — After referral to Columbia's outpatient pulmonary rehabilitation (PR) program, participants randomized to the Wait-List control group will be put on a PR wait list (usual care). In Phase II, all participants will receive PR of 1-hour sessions, twice per week for 10 weeks. Traditional outpatient PR: Group exercise training (ET) combined with pursed lips breathing (PLB) training; 1:2 therapist to patient ratio. Home Program: Unmonitored walking exercise 1-2 days/week; no biofeedback monitoring. Coaching: Traditional monitoring and verbal cueing. Personnel: PT or EP. Frequency:
  1-hour sessions, twice per week for 10 weeks. Exercises: • ET of muscles of ambulation with exercise equipment, such as on a treadmill or cycle ergometer (30-min), plus 15-min strengthening and posture exercises; O2 supplementation as needed. No breathing biofeedback. • PLB instruction only during exercise training. Education: Verbal and written information.
  Arms: Wait-List Control

SUMMARY:
This pilot study is part of a phased approach to refine, optimize, and test the feasibility of CALM Breathing. Preliminary participant feedback from the Capnography-Assisted Respiratory Therapy (CART) study was applied to adapt and design CALM Breathing (including its dose, schedule, delivery, and home program). This pilot builds on initial lessons learned and identifies intervention areas still needing greater development to assure the success of a future large trial, targeting a subpopulation at risk, that is, those with COPD and anxiety sensitivity.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate an experimental breathing therapy for adults with chronic obstructive pulmonary disease (COPD) called Capnography-Assisted Learned, Monitored (CALM) Breathing. CALM Breathing is an experimental therapy that uses exercises combined with breathing feedback. CALM Breathing promotes self-regulated breathing to relieve symptoms. In sessions, biofeedback of breathing is predominately provided by two devices that are cleared by the Food and Drug Administration (FDA) to measure carbon dioxide at the end of a breath and breathing rate. A capnograph uses tubing at the nose to evaluate levels of carbon dioxide and breathing rate from exhaled air and to display breathing patterns. A pulse oximeter for home use also evaluates breathing rate at the fingertip with a sensor that detects blood flow changes. The investigators are studying CALM Breathing to see if it can relieve shortness of breath and other symptoms; reduce stress; and improve quality of life and exercise tolerance in adults with COPD. The investigators are planning to recruit up to approximately 65 subjects with COPD at Columbia University Irving Medical Center. Participants will be assigned by chance into one of two treatment groups: 1) CALM Breathing or Usual Care (Waitlist). Participants will have an equal chance of being assigned to either group. CALM Breathing is a 4-week therapy program that uses breathing exercises with biofeedback to reduce shortness of breath and other symptoms related to COPD. Biofeedback uses sensors to give information about breathing pattern and airflow to help participants better self-regulate their breathing. Participants assigned by chance to CALM Breathing, will participate in eight breathing therapy sessions, provided twice per week; each session will each take approximately 1-hour. All participants will receive 16-20 standard care pulmonary rehabilitation sessions beginning at approximately week 6-10. Participants will complete three study evaluation visits (at baseline, ~6 weeks, and at a 3-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* be adult males or females
* have a diagnosis of COPD as defined by FEV1/FVC of < 0.70 on spirometry testing or as shown on a chest computed tomography (CT)
* receive standard care of pharmacotherapy with bronchodilators (e.g. long-acting beta-agonists, LABAs, or long-acting muscarinic antagonists, or LAMAs) as prescribed by their physician
* are in stable medical condition as determined by pulmonary rehabilitation physician (i.e., not in need of acute higher level of care such as hospitalization)
* have dyspnea [as documented in their medical record or based on self-report; e.g., ≥1 on modified Medical Research Council questionnaire (mMRC) dyspnea; or ≥2 dyspnea score on item: "Over the last 4 weeks, I have had shortness of breath: almost every day = 4, several days a week = 3, a few days a month = 2, only with lung/respiratory infections = 1, not at all = 0; or "yes" response of binary presence of dyspnea-related avoidance of activities: "Have you avoided any activities due to shortness of breath?")]
* have elevated dyspnea-related anxiety symptoms:

  * DMQ-CAT dyspnea anxiety score ≤50; or
  * DMQ-CAT activity avoidance ≤50;
  * VAS dyspnea anxiety scale score of ≥20, administered with 6-minute walk test;
  * ASI-16: item #10, "It scares me when I become short of breath (at least "some");
* require ≤ 24 hours per day of supplemental oxygen
* Mini-Mental State Examination score ≥24
* speak, read, and write English
* are stably medicated for at least 4 weeks prior to study entry with long-acting anti-anxiety medication (e.g., selective serotonin reuptake inhibitors, SSRIs, and serotonin norepinephrine reuptake inhibitors, SNRIs), benzodiazepines, or cannabis if prescribed, with no plans to change psychotropic medication dose
* have not received any pulmonary rehabilitation training in the past 12 months.

Exclusion Criteria:

* are not eligible for pulmonary rehabilitation
* are actively being treated for cancer
* have morbid obesity (Body Mass Index (BMI) > 40)
* have hypercapnia of ETCO2 > 50 mmHg at rest
* have a musculoskeletal disorder severe enough to interfere with walking or ability to exercise or have neuromuscular disease
* have had a seizure in the past 3 months
* reside in an acute hospital, sub-acute care, assisted living, or nursing home
* are active smokers
* are pregnant
* have any clinically significant cardiac disease or any electrocardiogram (ECG) abnormality obtained during the screening, which in the opinion of the investigator may put the patient at risk or interfere with study assessments
* have low literacy as indicated by scores of 4 or 5 ("often" and "always") on the Single Item Literacy Screener (SILS) that asks, "How often do you need to have someone help you when you read instructions, pamphlets, or other written material from your doctor or pharmacy?"
* have a diagnosis or medical history of schizophrenia, psychotic disorders, or bipolar disorder as diagnosed by study psychologist
* have alcohol or substance abuse or dependence within the past 6 months as evaluated by study psychologist
* have serious suicidal risk (suicidal ideation or suicidal behaviors within the past year) as defined by a score of >1 on psychologist interview-administered Clinician Suicide Assessment Checklist, which is a Modified Columbia-Suicide Severity Rating Scale-CSSRS
* Take prescribed opioids ≥50 MME (morphine mg equivalents) per day. A dosage threshold of ≥50 MME significantly increases the risk of fatal respiratory depression and necessitates additional precautions. Participants' opioid medication dose will be confirmed by their prescribing physician (e.g., their primary care or pain management doctor).
* Actively take both prescribed opioids and benzodiazepines. Combining benzodiazepines and opioids significantly increases the risk of respiratory failure in patients with chronic obstructive pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Norweg, PhD, OTR, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - New York University Grossman School of Medicine, New York, New York
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with Columbia University. Requests may be directed to the Principal Investigator (PI). The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements
Access Criteria: Requests may be directed to the PI.

REFERENCES:
- [Derived] Norweg A, Oh C, DiMango A, Hofferber B, Spinner M, Stavrolakes K, Pavol M, Lindenauer P, Murphy CG, Simon NM. Mind the Breath: Feasibility of Capnography-Assisted Learned Monitored (CALM) Breathing for Dyspnea Treatment. J Cardiopulm Rehabil Prev. 2025 Mar 1;45(2):118-131. doi: 10.1097/HCR.0000000000000939. Epub 2025 Feb 13. PMID 39976559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CALM Breathing | Wait-List Control
Started | 20 | 22
Randomized | 20 | 22
Started Pulmonary Rehab | 11 | 18
Completed (Refers to the completion of the study and not the pulmonary rehab.) | 9 | 19
Not Completed | 11 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CALM Breathing | Wait-List Control | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (7) | 70 (12) | 71 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 14 | 18 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Supplemental Oxygen (home use) [Count of Participants; unit: Participants] | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Attendance Rate of CALM Breathing Treatment Sessions
Description: Attendance rate will be measured from the total number of sessions completed out of the 8 total.
Time Frame: 4 weeks
Population: This outcome measure is only measuring attendance for individuals who received the CALM breathing intervention.
Measure: Mean (Full Range); unit: percentage of completed sessions
Arm/Group | CALM Breathing
Number analyzed (Participants) | 19
percentage of completed sessions | 84.2 [0 to 100]

2. Primary Outcome: Drop-Out Rate
Description: The drop-out rate will be calculated from the total number of participants who drop-out from receiving the CALM Breathing therapy.
Time Frame: 3 months
Population: This outcome measure is only looking to measure the drop-out rate for the CALM Breathing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | CALM Breathing
Number analyzed (Participants) | 19
Participants | 1

3. Primary Outcome: CALM Breathing Satisfaction Rating
Description: The acceptability of the CALM Breathing therapy will be evaluated based on mixed methods data collected from CALM Breathing satisfaction ratings.
  Participants were asked item 8 of FACIT ("how do rate this treatment overall?"), which was rated from 0 to 4 (0 = "poor" and 4 = "excellent") in which higher scores indicate more satisfaction (better outcome).
Time Frame: 4 weeks
Population: Only data from the 17 participants who completed the satisfaction questionnaire from the CALM Breathing arm was collected and analyzed.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | CALM Breathing
Number analyzed (Participants) | 17
score on a scale | 2 [0 to 4]

4. Secondary Outcome: Chronic Respiratory Disease Questionnaire (CRQ) Score
Description: This questionnaire measures the impact of chronic obstructive pulmonary disease (COPD) on a person's life. It consists of 20 items across 4 domains (dyspnea, fatigue, emotional function, and master). Items are on a 7-point Likert scale (1 - 7) and are scored from 1 (most severe) to 7 (no impairment) (better outcome). For this trial, questions 4a- 4e are included which is the dyspnea domain. The 5 scores are summated and divided by the number of items. The range is 1-7. Higher scores indicate better outcomes.
Time Frame: Baseline, 4 weeks, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 4.63 (1.5) | 4.06 (1.42)
  4 weeks | 5.24 (1.26) | 4.19 (1.25)
  3 months | 4.94 (1.45) | 4.31 (1.60)

5. Secondary Outcome: Dyspnea Management Questionnaire Computer Adaptive Test (DMQ-CAT) Score
Description: The DMQ-CAT is a 71-item questionnaire that measures dyspnea anxiety. Raw scores range from 0 (low) to 6 (high). These raw scores are converted into T-scores with a mean score of 50 and a standard deviation of ±10. The full range of T-scores is 0 to 100 for DMQ-CAT Self-Efficacy, DMQ-CAT Intensity and DMQ-CAT Anxiety scales. The DMQ-CAT software automatically scores these scales. Higher scores indicate better outcomes.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
T-score
  DMQ-CAT Self-Efficacy | 54.9 (6.1) | 53 (7)
  DMQ-CAT Intensity | 57 (8) | 54 (10)
  DMQ-Anxiety | 58 (7) | 52.1 (6)

6. Secondary Outcome: Dyspnea Management Questionnaire Computer Adaptive Test (DMQ-CAT) Score
Description: The DMQ-CAT is a 71-item questionnaire that measures dyspnea anxiety. Raw scores range from 0 (low) to 6 (high). These raw scores are converted into T-scores with a mean score of 50 and a standard deviation of ±10. The full range of T-scores is 0 to 100 for DMQ-CAT Self-Efficacy, DMQ-CAT Intensity and DMQ-CAT Anxiety scales. The DQM-CAT software automatically scores these scales. Higher scores indicate better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
T-score
  DMQ-CAT Self-Efficacy | 54.9 (5.8) | 54.0 (8.0)
  DMQ-CAT Intensity | 55.0 (10.0) | 53.0 (12.0)
  DMQ-Anxiety | 57 (8) | 52.7 (6)

7. Secondary Outcome: Modified Borg Scale Score
Description: The Modified Borg Scale is most commonly used to assess symptoms of breathlessness. On the 11-item scale, a score of 0 indicates "No Exertion" and a score of 10 indicates "Maximal" exertion (10-point scale). The full range is 0-10 for Borg-Dyspnea and Borg-Fatigue. Higher scores indicate worse outcomes (i.e. more exertion).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
score on a scale
  Borg Dyspnea | 4 (2) | 5 (4)
  Borg Fatigue | 3 (3) | 5 (4)

8. Secondary Outcome: Modified Borg Scale Score
Description: as for outcome 7
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
score on a scale
  Borg Dyspnea | 3 (2) | 5 (2)
  Borg Fatigue | 2 (3) | 4 (3)

9. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7) Score
Description: The General Anxiety Disorder-7 is a 7-item screening tool and symptom severity measure for the four most common anxiety disorders. This is calculated by assigning scores of 0 ("not at all"), 1 ("several days'), 2 ("more than half the days"), or 3 ("nearly every day"). GAD-7 total score for the seven items ranges from 0 to 21. Higher scores indicate worse outcomes (i.e. greater anxiety).
Time Frame: 3 months
Population: Data was not collected.
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Perceived Stress Scale Score (PSS)
Description: The PSS is a 10-item classic stress assessment instrument. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: Baseline, 4 weeks, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 12 (9) | 18 (7)
  4 weeks | 13 (9) | 21 (8)
  3 months | 10 (8) | 19 (7)

11. Secondary Outcome: 6 Mile Walking Distance Score (6MWT)
Description: This is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Time Frame: Baseline, 4 weeks, 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
meters
  Baseline | 304 (86) | 341 (109)
  4 weeks | 283 (106) | 319 (121)
  3 months | 295 (109) | 369 (94)

12. Secondary Outcome: Physical Activity Scale for the Elderly (PASE)
Description: This 12-item questionnaire uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity.
Time Frame: 3 months
Population: Data was not collected for this analysis.
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in COPD Assessment Test (CAT) Score
Description: The CAT quantifies the impact of COPD symptoms on patients' overall health. Participants assign a score ranging from 0 to 5 for each of the 8 areas. A score of 0 means there is no impairment in that area. A score of 5 means severe impairment. The overall score will range from 0 to 40. The score is a composite score.
Time Frame: 4 weeks, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
score on a scale
  Change from Baseline to 4 weeks | 1 (37) | 19 (5)
  Change from Baseline to 3 months | -6 (47) | 7 (35)

14. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-24).
Description: This is a 10-item tool used to measure patient-reported outcomes (PROs) relevant across common medical conditions. The response options are presented as a 5-point rating scale, with higher scores indicating a healthier patient (better outcome). Scores are standardized to the general population using the "T-Score", with the average T-score for the US population is 50 points, with a SD of 10 points. This applies to PROMIS Social, PROMIS Fatigue, PROMIS Physical, and PROMIS Sleep Disturbance.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
T-score
  PROMIS Social | 52 (10) | 45 (11)
  PROMIS Fatigue | 48 (12) | 59 (12)
  PROMIS Physical | 40.1 (6.6) | 36 (7)
  PROMIS Sleep Disturbance | 50.9 (6.9) | 54.7 (6.4)

15. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-24).
Description: as for outcome 14
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
T-score
  PROMIS Social | 52 (11) | 45 (9)
  PROMIS Fatigue | 52 (12) | 59 (10)
  PROMIS Physical | 39.4 (7.2) | 38 (7)
  PROMIS Sleep Disturbance | 51.3 (6.6) | 54.4 (5.5)

16. Secondary Outcome: End-tidal CO2
Description: This measures the partial pressure of CO2 at the end of an exhaled breath.
Time Frame: Baseline, 4 weeks, 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
mmHg
  Baseline | 30 (7) | 32.5 (5.4)
  4 weeks | 34 (8) | 31.1 (6.0)
  3 months | 31 (6) | 29.8 (3.7)

17. Secondary Outcome: Patient Activation Measure (PAM) Score
Description: Pulmonary Rehabilitation Engagement will be measured using the Patient Activation Measure (PAM), which is a 10 or 13 item questionnaire that measures patients on a 0-100 scale and can segment patients into one of four activation levels along an empirically derived continuum. Each activation level reveals insight into an array of health-related characteristics, including attitudes, motivators, behaviors, and outcomes. A higher score indicates a better outcome.
Time Frame: Baseline, 4 weeks, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 45 (5) | 43 (5)
  4 weeks | 45 (6) | 42 (6)
  3 months | 46 (5) | 44 (5)

18. Other Pre Specified Outcome: Self-Evaluation of Breathing Questionnaire (SEBQ) Score
Description: The SEBQ contains 12 items and assesses the patient's perception of their breathing difficulties and gives an insight into the effort of breathing and the feeling of air hunger. Responses to these items are on a 4-point Likert scale: (0) never/not true at all; (1) occasionally/a bit true; (2) frequently-mostly true; and, (3) very frequently/very true. SEBQ scores for sum of the original items ranged from 0 to 36, with a lower total indicating a better outcome.
Time Frame: Baseline, 4 weeks, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CALM Breathing | Wait-List Control
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 12 (8) | 19 (7)
  4 weeks | 11 (9) | 17 (6)
  3 months | 11 (9) | 17 (8)

ADVERSE EVENTS:
Time Frame: AE data was collected over 3 months from baseline or until the participants completed/withdrew from the study.
Groups:
- All Participants: All AEs that occurred for any study participant was recorded but not stratified per arm. AEs were not collected per arm and therefore stratified data is not available.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 5/42
Other Adverse Events (participants affected / at risk) | 11/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=42)
Chest Tightness (Cardiac disorders) | 1 (1) — 1 hospitalization due to chest tightness.
Hospitalization due to Missed Hemodialysis (Renal and urinary disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (2) — 2 hospitalizations due to pulmonary edema.
COVID-19 Infection (Infections and infestations) | 2 (2) — 2 hospitalizations due to COVID-19 infection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=42)
Stomach Flu (Infections and infestations) | 1 (1)
Anxiety (Social circumstances) | 1 (1) — Anxiety was related to pending eviction from apartment.
COPD Requiring Modified Treatment (Respiratory, thoracic and mediastinal disorders) | 6 (6) — Increased antibiotic and steroid use for COPD symptom management
UTI (Infections and infestations) | 1 (1) — UTI requiring antibiotic treatment
Sleepiness (General disorders) | 1 (1)
Fall (outdoors) (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT04786184/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT04786184/SAP_001.pdf
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT04786184/ICF_002.pdf